CLINICAL TRIAL: NCT02561598
Title: A Case Control Study of Patients With Diagnosis of Malignant Hyperthermia
Status: Withdrawn | Type: Observational
Why Stopped: Research Staffing issues
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-2884
Record Dates: First submitted 2015-07-27; First posted 2015-09-28 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Malignant Hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples from other approved projects will be used from both malignant hyperthermia cases and controls.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malignant Hyperthermia: Samples from persons who have a malignant hyperthermia diagnosis.
- Controls: Children who participated in pharmacogenetic research and had exposure to malignant hyperthermia triggering agents.

SUMMARY:
The purpose of the study is to develop methods to identify predictors of Malignant Hyperthermia.

DETAILED DESCRIPTION:
The current study will use the combination of electronic medical records and genomic information in samples of persons who have exhibited signs of Malignant Hyperthermia (MH) or have family history or high risk of MH to see if risk factors can be identified. These will be compared with control samples of children who have been exposed to the same agents which could induce MH, yet showed no signs of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Malignant hyperthermia cases: Diagnosis of malignant hyperthermia
* Control cases: children who participated

Exclusion Criteria:

* Not meeting the inclusion criteria stated above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases are selected from the medical records at Cincinnati Children's Hospital Medical Center who have a current malignant hyperthermia diagnosis. Control cases are selected based on previous participation in pharmacogenetic research and had exposure to agents known to trigger malignant hyperthermic episodes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Number of clinical manifestations of malignant hyperthermia | Within data collection period (3 years total).
  Incidence of clinical manifestations of MH will be compared among patients with a history of MH to controls (no diagnosis of MH).

SECONDARY OUTCOMES:
number of Genetic indications for malignant hyperthermia | Within data collection period (3 years total).
  genetic indications for malignant hyperthermia will be compared between control subjects and subjects with a diagnosis of MH

CONTACTS AND LOCATIONS:
Overall Officials: John McAuliffe, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States